CLINICAL TRIAL: NCT02018692
Title: The Effect of Oral Administration of 9-cis β Carotene Rich Powder of the Alga Dunaliella Bardawil on Visual Functions in Adolescent Patients With Retinitis Pigmentosa
Brief Title: The Effect of Oral Administration of 9-cis Rich Powder of the Alga Dunaliella Bardawil on Visual Functions in Adolescent Patients With Retinitis Pigmentosa
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Director, Electrophysiology Clinic, Goldschleger Eye Research Institute, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-13-9579-YR-CTIL
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alga Dunaliella Bardawil 9-cis beta Carotene Rich Powder (Experimental): 15 patients will first receive the capsules containing the alga Dunaliella Bardawil 9-cis beta-Carotene rich powder (5mg/Kg) for 24 weeks. After 24 weeks of washout period they will receive capsule containing placebo (Starch) for 24 weeks.
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil powder; Dietary Supplement: Placebo:Starch
- Placebo (Starch) (Placebo Comparator): The other 15 Patients will receive first the placebo (Starch) capsules for 24 weeks. After 24 weeks of washout period they will receive capsules containing the alga Dunaliella Bardawil 9-cis beta-Carotene rich powder .
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil powder; Dietary Supplement: Placebo:Starch

INTERVENTIONS:
Dietary Supplement: Alga Dunaliella Bardawil powder — 9 cis beta carotene rich Alga Dunaliella Bardawil powder
Dietary Supplement: Placebo:Starch — Starch powder

SUMMARY:
The aim of this study is to determine whether 9-cis-beta Caroten rich D. Brdawiil extract is effective in the treatment of retinitis pigmentosa in adolescent patients.

DETAILED DESCRIPTION:
Retinitis pigmentosa is a genetically disease consisting of progressive retinal degeneration starting in the rods. Its prevalence is 1:4000 people and is the fourth most common blinding disease in Israel in 2004 [7% of all blindness]. The investigators treated a non-progressive form of the disease [Fundus Albipunctatus] by oral therapy of the food supplement made from alga Dunaliella Bardawil composed of approximately 50% 9-cis β-carotene.

The 9-cis β -carotene has been shown to be a precursor of 9-cis retinoic acid both in-vitro in human intestinal mucosa and in-vivo in a ferret, perfused with 9-cis b-carotene. The night vision, as measured objectively by electroretinography (ERG) more than doubled in six patients tested following treatment. The visual field was also improved significantly. In a more recent study the investigators treated 29 retinitis pigmentosa patients with the 9-cis b Carotene algae Dunaliella Bardawil in a double masked placebo control cross over trial. Significant improvement in retinal function was recorded in 34% of the patients.

As a natural extension of this study we will perform a double-masked, randomized, crossover, placebo-controlled study for adolescent patients. Longer treatment duration will be tested: a 24 week treatment with either the 9-cis β-carotene-rich capsules or placebo followed by an additional a 24 week treatment with the other capsules and a wash-out period of 24 weeks between this two type of treatments. We predict that with this study design a maximal/increased therapeutic effect as well as efficient washout will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Adolescent 12-18 years old.
* Electroretinogram (ERG) responses compatible with the diagnosis of Retinitis Pigmentosa

Exclusion Criteria:

* Currently a smoker
* Current use of vitamin A/ β-carotene supplements
* Active arterial disease within 3 months prior to enrolment in the study, e.g. unstable angina, myocardial infarction, transient ischemic attack, stroke, coronary artery bypass graft surgery
* History of malignancy, excepting basal or squamous cell skin carcinoma
* Females who are pregnant, or breast feeding, or are premenopausal but not using chemical or mechanical contraception
* Uncontrolled hypertension, defined either as resting diastolic blood pressure >95 mmHg (taken from the mean of 3 readings) or as resting systolic blood pressure >180 mmHg
* History of alcohol abuse or drug abuse or both
* Intention to engage in vigorous exercise or an aggressive diet regimen
* Uncontrolled endocrine or metabolic disease
* Participation in another investigational drug study within 4 weeks prior to enrolment
* Serious or unstable medical or psychological condition which, in the opinion of the PI, would compromise the subject's safety or successful participation in the study
* Initiation of hormone replacement therapy or oral contraceptive therapy within 3 months prior to enrolment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean binocular maximal scotopic electroretinogram b-wave response | up to weeks 72
  Using the protocol of the International Society for Clinical Electrophysiology of Vision and the "UTAS 3000" system (LKC Technologies, Gaithersburg, MD), full-field electroretinographic responses will be recorded from both eyes of each patient. For scotopic conditions, maximal ERG b-wave responses will be recorded following 30 minutes of dark adaptation.

SECONDARY OUTCOMES:
The area within the Dark adapted chromatic Goldamann Visual field in isopters in cm2 | On weeks 0, 24, 48, 72
  Kinetic visual field for chromatic stimuli will be recorded in both eyes after 30 minutes of dark adaptation. Area of vision within the isopter will be measured by software in cm2.
The area within Goldamann Visual field in isopters in cm2 | On weeks 0, 24, 48, 72
  Kinetic visual field will be recorded in both eyes. Area of vision within the isopter will be measured by software in cm2.
Mean binocular maximal photopic electroretinogram b-wave response | On weeks 0, 24, 48, 72
  Using the protocol of the International Society for Clinical Electrophysiology of Vision and the UTAS 3000 system (LKC Technologies, Gaithersburg, MD), full-field photopic electroretinographic responses will be recorded from both eyes of each patient.
Best-corrected visual acuity (EDTRS) | On weeks 0, 24, 48, 72
Objective visual field by chromatic multifocal pupillometer | On weeks 0,24,48,72

CONTACTS AND LOCATIONS:
Overall Officials: Ygal Rotenstreich, MD, Principal Investigator — Goldschleger Eye Research Institute, Sheba Medical Center, Tel Hashomer
Locations (1):
- Goldschleger Eye Research Institute, Sheba Medical Center,, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotenstreich Y, Belkin M, Sadetzki S, Chetrit A, Ferman-Attar G, Sher I, Harari A, Shaish A, Harats D. Treatment with 9-cis beta-carotene-rich powder in patients with retinitis pigmentosa: a randomized crossover trial. JAMA Ophthalmol. 2013 Aug;131(8):985-92. doi: 10.1001/jamaophthalmol.2013.147. PMID 23700011
- [Background] Skaat A, Sher I, Kolker A, Elyasiv S, Rosenfeld E, Mhajna M, Melamed S, Belkin M, Rotenstreich Y. Pupillometer-based objective chromatic perimetry in normal eyes and patients with retinal photoreceptor dystrophies. Invest Ophthalmol Vis Sci. 2013 Apr 17;54(4):2761-70. doi: 10.1167/iovs.12-11127. PMID 23482470
- [Background] Rotenstreich Y, Harats D, Shaish A, Pras E, Belkin M. Treatment of a retinal dystrophy, fundus albipunctatus, with oral 9-cis-beta-carotene. Br J Ophthalmol. 2010 May;94(5):616-21. doi: 10.1136/bjo.2009.167049. Epub 2009 Dec 2. PMID 19955196
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764